CLINICAL TRIAL: NCT06516783
Title: Evaluation of the Effectiveness and Safety of Blue Light Emitted by LED Lamps Using the PHLECS Device in the Treatment of Inflammatory Skin Diseases
Brief Title: Blue Light in the Treatment of Inflammatory Skin Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Magdalena Sadowska, MD, Medical University of Lodz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMED-RNN/223/20/KE
Record Dates: First submitted 2024-06-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Atopic Dermatitis; Psoriasis Vulgaris; Eczema; Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with psoriasis, atopic dermatitis, eczema and chronic pruritus (Experimental): The study is scheduled for a maximum of 60 irradiations of blue light (maximum 3 cycles of 20 irradiations each). Phototherapeutic light will be administered for 15 minutes to each side of the body of the patient (30 minutes in total), 3-5 times per week.
  • Device Full Body Blue GEN 1.0 device (built by PHLECS B.V.) with European Community (EC) Certificate (number 2238613CE01) is used in the study. The device provides phototherapeutic light through light panel with treatment Light Emitting Diodes - LEDs (wavelength 453 nm, irradiance 40mW/cm2; dose 36J for 15min treatment) to one side of the body of the patient who is lying flat on an examination bed
  Interventions: Device: Full Body Blue GEN 1.0 device

INTERVENTIONS:
Device: Full Body Blue GEN 1.0 device — Full body blue irradiation in the treatment of inflammatory skin diseases and chronic pruritus

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of full-body blue light irradiations in the treatment of inflammatory skin diseases (atopic dermatitis, psoriasis, eczema) and chronic pruritus in adult and pediatric populations.

The main questions it aims to answer are:

* If blue light irradiations have an impact on the improvement in skin condition
* If blue light irradiations affect the patients' quality of life
* If blue light irradiations decrease pruritus

Participants will:

* Be administered phototherapeutic blue light (453 nm) for 15 minutes to each side of the body (30 minutes in total), 3-5 times per week. The study is scheduled for a maximum of 60 irradiations of blue light.
* Complete the Dermatology Life Quality Index questionnaire and a 10-item pruritus severity scale
* Be assessed using dermatologic scales
* Have blood samples collected

DETAILED DESCRIPTION:
After giving written, informed consent, skin examination will be performed (including photo documentation) and each patient will have skin phototype assessed according to Fitzpatrick's scale. A detailed medical history will be collected. In addition, patients will complete the Dermatology Life Quality Index (DLQI) questionnaire and 10-item pruritus severity scale. Clinical assessment will be performed depending on the disease:

PASI, PGA, VAS, 10-item Pruritus Severity Scale - psoriasis vulgaris;

IGA, VAS, 10-item Pruritus Severity Scale - eczema;

SCORAD, EASI, VAS, 10-item Pruritus Severity Scale - atopic dermatitis;

VAS, 10-item Pruritus Severity Scale - chronic pruritus.

On day 0, before the start of the treatment blood samples will be collected. Optionally, with additional consent, a skin biopsy will be taken. The study is scheduled for a maximum of 60 irradiations of blue light (maximum 3 cycles of 20 irradiations each). Phototherapeutic light (wavelength 453 nm, irradiance 40mW/cm2; dose 36J for 15min treatment) will be administered for 15 minutes to each side of the body of the patient (30 minutes in total), 3-5 times per week using the PHLECS Full Body Blue device (with European Community Certificate number 2238613CE01).

Visits schedule:

Visit 1 - First irradiation;

Visit 2 - evaluation of the effectiveness and safety after 10 sessions of blue light phototherapy, blood sample collection;

Visit 3 - evaluation of the effectiveness and safety after 20 sessions of blue light phototherapy (= after the first cycle of irradiation), Blood sample collection;

Visit 4 - evaluation of the effectiveness and safety after 30 sessions of blue light phototherapy, Blood sample collection;

Visit 5 - evaluation of the effectiveness and safety after 40 sessions of blue light phototherapy (= after the second cycle of irradiation), Blood sample collection;

Visit 6 - evaluation of the effectiveness and safety after 50 sessions of blue light phototherapy, Blood sample collection;

Visit 7 - end of treatment visit - after 60 sessions of blue light phototherapy (= after the third radiation cycle), during which we will re-evaluate the condition of the skin, quality of life, safety of the device used and blood samples will be taken. Optionally, with additional consent, a skin biopsy will be taken. If, for any reason, the study is terminated earlier or if the skin lesions have completely disappeared before 60 irradiations - the end of treatment visit will take place earlier;

Visit 8 - assessment of the clinical condition 4 weeks after the cessation of therapy.

During blue light therapy, follow-up visits will be performed to assess the safety and effectiveness of the device. At the last control visit (end of treatment visit) the same parameters will be assessed as during the first one. In the case of remission of skin lesions earlier than envisaged in the study protocol, the end of treatment visit will take place earlier. Photographic documentation will be carried out at each visit. During the treatment patients will be allowed to use emollients. Statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in a medical experiment
* Age above 8 years of age
* Diagnosis of psoriasis / eczema / atopic dermatitis
* Chronic pruritus (lasting more than 6 weeks)
* Good general health (no history of other clinically significant diseases according to the doctor's assessment)
* A patient who is able to understand the information related to the experiment, meet the requirements contained in the protocol of the experiment, who undertakes to strictly follow medical recommendations and appear on time for visits.

Exclusion Criteria:

* Patients with known hypersensitivity to ultraviolet or blue radiation
* Age under 8 years of age
* Women who are pregnant, breastfeeding or planning to become pregnant during the experiment
* Patients who participated in another experiment / clinical trial within 30 days prior to inclusion in the experiment
* Patients unwilling or unable to respect the requirements of the experiment
* Patients with skin diseases other than inflammatory skin diseases or chronic pruritus
* Planned hospitalizations or surgical procedures during the medical experiment
* Patients using medications with proven phototoxic effect
* Diastolic blood pressure> 95mmHg and <65mmHg
* Patients with congenital or acquired immune disorders
* Patients with a history or at the time of the examination diagnosed with a malignant skin cancer, severe actinic keratosis or dysplastic moles
* Patients diagnosed with genophotodermatosis, increasing the risk of skin cancers, including xeroderma pigmentosum, Cockayne's syndrome, Bloom's syndrome)
* Patients addicted to alcohol / drugs in the last 12 months

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Statistically significant change in PASI (Psoriasis Area Severity Index) score of the patients after blue light irradiation | From the date of the first irradiation (visit 1) until the cessation of therapy, up to 25 weeks. In case of earlier cessation of therapy, the evaluation will be conducted at the last visit and then 4 weeks after the cessation of therapy.
  Statistically significant (p <0.05) change in skin condition of the patients after blue light irradiations using:
  PASI - Psoriasis Area Severity Index (0-72 points; higher scores mean a worse outcome) in patients with psoriasis vulgaris
Statistically significant change in PGA (Physician's Global Assessment) score of the patients after blue light irradiation | From the date of the first irradiation (visit 1) until the cessation of therapy, up to 25 weeks. In case of earlier cessation of therapy, the evaluation will be conducted at the last visit and then 4 weeks after the cessation of therapy.
  Statistically significant (p <0.05) change in skin condition of the patients after blue light irradiation using:
  PGA - Physician's Global Assessment (0-5 points; higher scores mean a worse outcome) in patients with psoriasis vulgaris
Statistically significant change in VAS (Visual Analogue Scale) score of the patients after blue light irradiation | From the date of the first irradiation (visit 1) until the cessation of therapy, up to 25 weeks. In case of earlier cessation of therapy, the evaluation will be conducted at the last visit and then 4 weeks after the cessation of therapy.
  Statistically significant (p <0.05) change in skin condition of the patients after blue light irradiation using:
  VAS - Visual Analogue Scale (0-10 points; higher scores mean a worse outcome) in patients with psoriasis vulgaris, atopic dermatitis, eczema and chronic pruritus
Statistically significant change in 10-item Pruritus Severity Scale score of the patients after blue light irradiation | From the date of the first irradiation (visit 1) until the cessation of therapy, up to 25 weeks. In case of earlier cessation of therapy, the evaluation will be conducted at the last visit and then 4 weeks after the cessation of therapy.
  Statistically significant (p <0.05) change in skin condition of the patients after blue light irradiation using:
  10-item Pruritus Severity Scale (3-20 points; higher scores mean a worse outcome) in patients with psoriasis vulgaris, atopic dermatitis, eczema and chronic pruritus
Statistically significant change in IGA (Investigators' Global Assessment) score of the patients after blue light irradiation | From the date of the first irradiation (visit 1) until the cessation of therapy, up to 25 weeks. In case of earlier cessation of therapy, the evaluation will be conducted at the last visit and then 4 weeks after the cessation of therapy.
  Statistically significant (p <0.05) change in skin condition of the patients after blue light irradiation using:
  IGA - Investigators' Global Assessment (0-5 points; higher scores mean a worse outcome) in patients with eczema
Statistically significant change in SCORAD (SCORing Atopic Dermatitis) score of the patients after blue light irradiation | From the date of the first irradiation (visit 1) until the cessation of therapy, up to 25 weeks. In case of earlier cessation of therapy, the evaluation will be conducted at the last visit and then 4 weeks after the cessation of therapy.
  Statistically significant (p <0.05) change in skin condition of the patients after blue light irradiation using:
  SCORAD - SCORing Atopic Dermatitis (0-103 points; higher scores mean a worse outcome) in patients with atopic dermatitis
Statistically significant change in EASI (Eczema Area Severity Index) score of the patients after blue light irradiation | From the date of the first irradiation (visit 1) until the cessation of therapy, up to 25 weeks. In case of earlier cessation of therapy, the evaluation will be conducted at the last visit and then 4 weeks after the cessation of therapy.
  Statistically significant (p <0.05) change in skin condition of the patients after blue light irradiation using:
  EASI - Eczema Area Severity Index (0-72 points; higher scores mean a worse outcome) in patients with atopic dermatitis
Statistically significant (p <0.05) change in DLQI (Dermatology Life Quality Index) | From the date of the first irradiation (visit 1) until the cessation of therapy, up to 25 weeks. In case of earlier cessation of therapy, the evaluation will be conducted at the last visit and then 4 weeks after the cessation of therapy.
  Statistically significant (p <0.05) change in DLQI (Dermatology Life Quality Index; 0-30 points; higher scores mean a worse outcome) after blue light irradiations in patients with psoriasis vulgaris, atopic dermatitis, eczema, chronic pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Sadowska, Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Dermatology, Pediatric Dermatology and Dermatological Oncology, Medical University of Lodz, Lodz, Poland

REFERENCES:
- [Derived] Sadowska M, Narbutt J, Nolberczak D, Ciazynska M, Skibinska M, Sobolewska-Sztychny D, Aubert D, Lesiak A. Prospective Clinical Study: Full-Body Blue Irradiation in the Treatment of Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2631-2643. doi: 10.1007/s13555-024-01248-3. Epub 2024 Aug 24. PMID 39180711

DOCUMENTS (1):
  • Study Protocol (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT06516783/Prot_000.pdf